CLINICAL TRIAL: NCT02638558
Title: Evaluation of the Impact of Direct Conversation With Patients in the Compliance With the "Split-dose" Regimen Preparation for Colonoscopy Scheduled in the First Part of the Morning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Alida Andrealli, MD, Valduce Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 04/2015
Record Dates: First submitted 2015-11-30; First posted 2015-12-23 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2015-12

CONDITIONS: Colonoscopy Preparation Acceptance

ARMS (2):
- written + oral explanation (Experimental): patients will undergo both written and oral explanation for preparation with split dose
  Interventions: Other: written + oral explanation
- written explanation (Experimental): patients will receive only a written explanation for preparation with split dose
  Interventions: Other: written explanation

INTERVENTIONS:
Other: written + oral explanation
  Arms: written + oral explanation
Other: written explanation
  Arms: written explanation

SUMMARY:
Split-dose cleansing regimens for colonoscopies, independently from the type of laxative used, are now recommended over full (one day)-dose regimens from all the major guidelines. It is wellknown that splitting the dose (half of the dose the night before and half the day of the colonoscopy) is safe and guarantees a better cleansing of the colon and thus a higher chance of identifying mucosal lesions. This is crucial both in terms of achieving a high-quality colonoscopy and in terms of time and money saved.

Still, there are some issues about compliance and tolerability with split-dose regimens. Two recent prospective works have shown that only a small number of patients (33%) chooses the split-dose regimen when the colonoscopy is scheduled before 10 a.m. and when patients are forced to used the split-dose, 1/7 did not comply with it, especially if the procedure is before 10 a.m. The most common concerns are about early wake-up, travel interruption and fear of incontinence. Both these papers state that strategies to reduce this noncompliance are needed.

The investigators aim to prove whether an "active action" (an oral explanation before the colonoscopy about why split-dose regimens are better) may improve patients' compliance in endoscopies scheduled in the early morning (from 8 to 10 a.m).

ELIGIBILITY:
Inclusion Criteria:

* every patient who needs a colonoscopy

Exclusion Criteria:

* incapacity in reading and/or in oral comprehension
* contraindications in drinking the preparation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2016-01; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
patients compliance in taking split-dose preparation in the early morning colonoscopies | 4 months